CLINICAL TRIAL: NCT05044910
Title: The Impact of Malnutrition on Immune Responses to Tuberculosis in Indian Children
Brief Title: The Impact of Malnutrition on Immune Responses to Tuberculosis
Acronym: TBMAM
Status: Active, not recruiting | Type: Observational
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: Institute of Child Health, Madras Medical College, Chennai (Unknown); Stanley Medical College (Other Government); Kanchi Kamakoti Childs Trust Hospital, Chennai, India (Unknown); Queen Mary University of London (Other); London School of Hygiene and Tropical Medicine (Other); DBT, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019037
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition, Child; Tuberculosis
Keywords: malnutrition; moderate acute malnutrition; immunology
MeSH Terms: conditions — Child Nutrition Disorders; Tuberculosis; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MAM children with TB disease
  Interventions: Dietary Supplement: Ready to Use supplementary food (RUSF)
- Wellnourished children with TB disease
- MAM children with latent TB infection
  Interventions: Dietary Supplement: Ready to Use supplementary food (RUSF)
- Well-nourished children with latent TB infection

INTERVENTIONS:
Dietary Supplement: Ready to Use supplementary food (RUSF) — Children with malnutrition will be given RUSF
  Groups: MAM children with TB disease; MAM children with latent TB infection

SUMMARY:
The aim of this study is to assess immune responses to Mtb in children with MAM compared to well-nourished children and to evaluate the impact of a nutrition intervention on these immune responses.

DETAILED DESCRIPTION:
Immune dysfunction in malnourished children is poorly characterised. The aim of this study is to assess immune responses to Mycobacterium tuberculosis (Mtb) in children with moderate acute malnutrition (MAM) compared to wellnourished children and to evaluate the impact of a nutrition intervention on these immune responses. Innate and adaptive immune responses to Mtb will be characterised in four groups: 1) MAM children with TB disease; 2) Wellnourished children with TB disease; 3) MAM children with latent TB infection; 4) Well-nourished children with latent TB infection. A range of assays to compare innate, adaptive and functional immune responses to TB between groups will be performed. Whether nutritional supplementation improves immune function in MAM children remains uncertain. Hence, children in all four groups will be followed up during 6 months of TB therapy/chemoprophylaxis. MAM children will receive 12 weeks of concomitant ready-to-use supplementary food, to evaluate longitudinal changes in innate and adaptive immune function, monocyte:lymphocyte ratio and mycobacterial growth inhibition. The results of this study will provide data to understand the reasons for infection susceptibility in malnourished children and provide a proof-of-concept that nutritional rehabilitation promotes immune rehabilitation. It will also provide a proof-of concept for use of nutritional supplementation as adjust therapy in TB disease

ELIGIBILITY:
Inclusion Criteria:

* Age 12-60 months
* HIV-negative
* BCG vaccinated
* Moderate acute malnutrition (WHZ -2 to -3 or MUAC 115 - 125mm ± HAZ <-2)
* TB disease
* Latent TB infection

Exclusion Criteria:

* Inclusion criteria not met
* Severe acute malnutrition (WHZ<-3; MUAC<115mm; bilateral oedema)
* Severe anaemia (Hb: <7g/dl)
* Chronic infection (HIV, hepatitis B or C)
* Chronic disease (e.g. Crohn's disease)
* Feeding problems (eg cerebral palsy) that prevent ingestion of RUSF
* Known nut allergy
* MDR TB disease and contacts of MDR TB adults

Ages: 12 Months to 60 Months | Sex: All
Age Groups: Child
Study Population: HIV negative, BCG vaccinated
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
IFNγ concentration | 6 months
  IFNγ concentration in supernatant after overnight incubation of whole blood with TB antigens

CONTACTS AND LOCATIONS:
Overall Officials: Aishwarya Venkataraman, MRCPCH, Principal Investigator — ICMR-NIRT
Locations (2):
- India (2):
  - Institute of Child Health, Chennai, Tamil Nadu
  - Government Stanley Medical College and Hospital, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No
Data will be shared according to ICMR rules and regulations after appropriate approvals

REFERENCES:
- [Derived] Venkataraman A, Shanmugam S, Balaji S, Mani K, Shanmugavel AK, Muthuramalingam K, Hissar S, Thiruvengadam K, Selladurai E, Smuk M, Hanna LE, Prendergast AJ. Comparison of two mycobacterial strains in performance of the whole blood mycobacterial growth inhibition assay in Indian children. Tuberculosis (Edinb). 2022 Dec;137:102255. doi: 10.1016/j.tube.2022.102255. Epub 2022 Aug 31. PMID 36252397